CLINICAL TRIAL: NCT02624505
Title: To Compare the Bronchoprotective Effects of the Test and Reference Metered Dose Inhalers (MDIs) Containing Albuterol Sulfate Using Methacholine Bronchoprovocation Challenge Testing in Stable Mild Asthma Patients.
Brief Title: Pharmacodynamic Bioequivalence of Metered Dose Inhalers of Albuterol Sulfate in Patients With Stable Mild Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: U-SS-M-AS312
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Product (Placebo Comparator): One actuation each from two different placebo Reference inhalation aerosols and one actuation each from two different placebo Test inhalation aerosols
  Interventions: Drug: Placebo
- 90 mcg Reference Product (Active Comparator): Drug : 90 mcg Reference Product One actuation each from the Reference inhalation aerosol and the placebo Reference inhalation aerosol and one actuation each from two different placebo Test inhalation aerosols
  Interventions: Drug: 90 mcg Reference Product
- 180 mcg Reference Product (Active Comparator): Drug: 180 mcg Reference Product One actuation each from two different Reference inhalation aerosols and one actuation each from two different placebo Test inhalation aerosols
  Interventions: Drug: 180 mcg Reference Product
- 90 mcg Test Product (Experimental): Drug: 90 mcg Test Product One actuation each from the Test inhalation aerosol and the placebo Test inhalation aerosol and one actuation each from two different placebo Reference inhalation aerosols
  Interventions: Drug: 90 mcg Test Product

INTERVENTIONS:
Drug: 90 mcg Reference Product — Drug: 90 mcg Reference Product
  Other Names: Albuterol
  Arms: 90 mcg Reference Product
Drug: 180 mcg Reference Product — Drug: 180 mcg of Reference Product
  Other Names: Albuetrol
  Arms: 180 mcg Reference Product
Drug: 90 mcg Test Product — Drug: 90 mcg of Test Product
  Other Names: Albuterol
  Arms: 90 mcg Test Product
Drug: Placebo — Placebo Product
  Arms: Placebo Product

SUMMARY:
The purpose of this study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product, using bronchoprovocation (methacholine challenge testing) in adult patients with stable mild asthma.

DETAILED DESCRIPTION:
This study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product in terms of FEV1 measured at different time-points, using bronchoprovocation (methacholine challenge testing) in adult patients with stable mild asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects (18-65 years of age)
* Forced Expiratory Volume in 1 second (FEV1) ≥ 80% of predicted. Airway responsiveness to methacholine demonstrated by a pre-albuterol dose (baseline) PC20 ≤ 8 mg/ml.
* Stable mild asthmatics based on National Asthma Education and Prevention Program (NAEPP) guidelines.
* Nonsmokers for at least 6 months prior to the study and a maximum smoking history of five pack-years (the equivalent of one pack per day for five years).
* Written informed consent.

Exclusion Criteria:

* Conditions which could alter airway reactivity to methacholine (e.g., pneumonia, upper respiratory tract infection, viral bronchitis and/or sinobronchitis) within six weeks prior to the screening visit.
* History of seasonal asthma exacerbations, in which case the patient should be studied outside of the relevant allergen season.
* History of a clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia.
* History of cystic fibrosis, bronchiectasis or other respiratory diseases other than Asthma
* Historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases
* Known intolerance or hypersensitivity or hypersensitivity to any component of the albuterol metered dose inhaler (MDI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Provocative Concentration of Methacholine Causing 20 % Fall (PC20) in FEV1(Forced Expiratory Volume in 1 second) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Abhyankar, Study Chair — Cipla Ltd.
Locations (1):
- Colorado Allergy and Asthma Centers, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Undecided